CLINICAL TRIAL: NCT02616016
Title: Magnetic Resonance-Guided High Intensity Focused Ultrasound for Palliation of Painful Skeletal Metastases in Children - A Pilot Study
Brief Title: MRI Guided HIFU for Palliation of Painful Skeletal Metastases in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We had challenges related to participant recruitment due to inclusion/exclusion criteria.
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, James Drake, Neurosurgeon, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000040604
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Bone Metastases; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI guided High Intensity Focused Ultrasound Treatment (Other): Intervention Group The interventional radiologist will locate the target tissue and mark the volume to be treated using MRI images.
  The operator starts the treatment and monitors the progress of the treatment with MR thermal and dose maps to ensure adherence to treatment plan.
  An individual treatment sonication will last approximately 30 seconds.
  Interventions: Device: MRI Guided High Intensity Focused Ultrasound

INTERVENTIONS:
Device: MRI Guided High Intensity Focused Ultrasound — Target treatment of bone metastases using High Intensity Focused Ultrasound

SUMMARY:
The Philips Sonalleve MR-HIFU system is expected to be effective in reducing pain intensity and/or reducing analgesic use in patients with painful uncomplicated bone metastases. No serious adverse effects are expected to result from this treatment.

DETAILED DESCRIPTION:
The objective of this study is to determine if MR-guided high intensity focused ultrasound (MR-HIFU) is an effective technique for alleviating the pain associated with bone metastases in paediatric cancer patients. This technique meant to be an adjunct therapy to the standard-of-care, which includes radiation therapy and chemotherapy. Safety of the technique will be assessed through evaluating non-targeted heating using MRI-based temperature mapping, and inspecting patients post-treatment for skin burns. or other signs of serious adverse events. Efficacy of the technique will be assessed by evaluating/recording patients observed pain, quality of life, and pain medication usage both before and up to 3 months following treatment.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent
* weight <140 kg (requirement to fit safely on top of the HIFU table and inside MRI
* any radiologic evidence of bone metastases from any solid tumor (neuroblastoma, osteosarcoma, soft tissue sarcoma, or any other solid tumor metastases).
* pain specifically at the site of interest (target lesion)
* pain score for target lesion >/ = 4 (indicating at least moderate pain) on an age-appropriate 0-10 point scale
* Target lesion in uncomplicated (ie no fracture / spinal cord compression /cauda equine syndrome/ soft tissue component)
* Available 3D MRI image of the target lesion (or be able to obtain one in a clinically feasible amount of time as part of the baseline investigational stage.)
* Proposed MR-HIFU treatment date >/= 2 weeks from most recent treatment of target tumour or systems chemotherapy
* Proposed MR-HIFU treatment date >/= 1 week after administration of steroids for pain flare

Exclusion Criteria:

* Unable to characterize pain specifically at the site of interest (target lesion).
* Pregnant / nursing females
* Target lesion is complicated (ie pressure of one fracture /spinal cord compression/cauda equine syndrome/soft tissue component)
* Target lesion < 1cm from nerve bundles/ bladder/bowel
* Target lesion in contact with hollow viscera
* Target lesion located in skull, spine (excluding sacrum which is allowed) or sternum.
* scar along proposed HIFU beam path.
* Orthopaedic implant along proposed HIIFU beam path or at site of target lesion.
* Active infection.
* Contradiction to general anesthesia or or gadolinium MRI contrast agent.
* Requirement for general anaesthesia for non -HIFU related MRI scans.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity scores from baseline as measured on pain diaries. | 2, 7, 14, 30 and 90 days following treatment
  As measured on the pain diaries before and at day 2, 7, 14, 30 and 90 days following treatment.

SECONDARY OUTCOMES:
Improved patient quality of life after MR-HIFU using a quality of life questionnaire. | 2, 7, 14, 30 and 90 days post treatment
  Using age appropriate quality of life questionnaire that involves interviewing patient and/or parent/guardian before and 2, 7, 14, 30 and 90 days post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: James M Drake, FRCSC,FACS, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada